CLINICAL TRIAL: NCT03642405
Title: Exploring the Effect of Methylphenidate and Antidepressants on Cardiac Repolarisation.
Brief Title: Drug-induced Repolarization ECG Changes
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Principal Investigator, Peter Marstrand, MD research fellow (Ph.D), Copenhagen University Hospital at Herlev
Other Study IDs: HerlevH01
Record Dates: First submitted 2018-08-16; First posted 2018-08-22 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2019-01

CONDITIONS: Long QT Syndrome; ADHD; Depression; Death; Death, Sudden, Cardiac; Romano-Ward Syndrome; Pathologic Processes; Heart Arrest; Electrocardiogram: Electrical Alternans; Heart Diseases; Cardiovascular Diseases; Death, Sudden; Arrhythmias, Cardiac; Heart Defects, Congenital; Cardiovascular Abnormalities; Congenital Abnormalities; Genetic Disease; Genetic Syndrome; Qt Interval, Variation in; Psychiatric Disorder
MeSH Terms: conditions — Long QT Syndrome; Attention Deficit Disorder with Hyperactivity; Depression; Death; Death, Sudden, Cardiac; Romano-Ward Syndrome; Pathologic Processes; Heart Arrest; Heart Diseases; Cardiovascular Diseases; Death, Sudden; Arrhythmias, Cardiac; Heart Defects, Congenital; Cardiovascular Abnormalities; Congenital Abnormalities; Genetic Diseases, Inborn; Mental Disorders | interventions — Echocardiography; Blood Specimen Collection; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Methylphenidate-Group: The group is examined before and after intake of Methylphenidate
  Interventions: Diagnostic Test: Electrocardiogram examination; Diagnostic Test: Echocardiography; Procedure: Blood Samples; Behavioral: Questionnaire
- Methylphenidate and know QT-prolonging SSRI: The group is examined before and after intake of Methylphenidate
  Interventions: Diagnostic Test: Electrocardiogram examination; Diagnostic Test: Echocardiography; Procedure: Blood Samples; Behavioral: Questionnaire
- Methylphenidate and non-QT-prolonging SSRI: The group is examined before and after intake of Methylphenidate
  Interventions: Diagnostic Test: Electrocardiogram examination; Diagnostic Test: Echocardiography; Procedure: Blood Samples; Behavioral: Questionnaire

INTERVENTIONS:
Diagnostic Test: Electrocardiogram examination — 12-lead ECG monitored by Holter
Diagnostic Test: Echocardiography — Echocardiography in accordance to Danish Society of Cardiology
Procedure: Blood Samples — Blood Samples include, Genetic analysis, serum-Methylphenidate, serum-Citalopram. Sodium, Potassium, Magnesium, Calcium, Chloride, White-Blood-Count, Hemoglobin, C-reactive-Protein, Creatinine, Carbamide, aspartate aminotransferase (ASAT), alanine aminotransferase (ALAT), Glucose and pro-brain natriuretic peptide (Pro-BNP).
Behavioral: Questionnaire — Questionnaire regarding patients quality of life

SUMMARY:
Studies have shown that the risk of developing heart arrhythmias, is increased in patients receiving medication for Attention-deficit hyperactivity disorder (ADHD) and depression. The QT-interval on a electrocardiogram (ECG) is often used to assess the patients risk of developing heart arrhythmias. The QT-interval defines the hearts electrical resting period and a long interval is linked to an increased risk of developing heart arrhythmias. In this project the investigators wish to examine possible side-effects in patients receiving medication for ADHD and depression and their dynamic QT-interval changes, by analysing the ECG changes that occur during "Brisk Standing".

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Patients treated with Methylphenidate
* Patients treated with Methylphenidate and QT-prolonging SSRI
* Patients treated with Methylphenidate and a non QT-prolonging SSRI

Exclusion Criteria:

* Patients considered in an unstable phase in their psychiatric condition
* Patients that are not able to understand the information regarding the trial, or who are unable to cooperate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50 Patients treated with Methylphenidate 50 Patients treated with Methylphenidate and QT-prolonging SSRI 50 Patients treated with Methylphenidate and a non QT-prolonging SSRI
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-08-15 (Actual); Primary Completion 2019-09-03 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
ECG changes | Through study completion, an average of 1 year.
  The Primary Outcome assess whether there are changes on ECG, primary the QTc-interval, in participants receiving medication for ADHD and depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Herlev Hospital, Herlev, Denmark